CLINICAL TRIAL: NCT06895083
Title: Comparison of Self-ligating Mico One and Conventional MBT Brackets Regarding Alignment Efficiency and Pain Experience- a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shoaib Rahim (Other)
Collaborators: Foundation University Islamabad (Other)
Responsible Party: Sponsor-Investigator, Shoaib Rahim, Assistant professor, Foundation University Islamabad
Organization: Foundation University Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FF/FUMC/215-329Phy/23
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: alignment efficiency and pain experience
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a single-blind, randomized parallel-arm study with two arms. Participants will be randomly assigned to either receive self ligating brackets or conventional brackets regarding Alignment efficiency and pain experience.
Masking Description: Interventional or control group will be selected randomly through sealed envelope by an independent researcher not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional (No Intervention): Participants in this arm will conventional brackets
- Experimental (Experimental): Participants in this arm will self ligating brackets
  Interventions: Other: self ligating brackets

INTERVENTIONS:
Other: self ligating brackets — selfligating are new brackets
  Arms: Experimental

SUMMARY:
The rate of Orthodontic tooth movement affects the efficacy and time duration of the treatment. One of the key factors, during the initial alignment phase, is the amount of the force that the arch-wire applies to the dentition. The amount of the applied force and the rate of tooth movement are directly proportional to the frictional resistance between the arch wire and bracket. The quality and degree of resistance is related to the physical characteristics of the arch wire, bracket material, arch wire dimensions, and the type of arch wire ligation. The estimated rate of tooth movement is about 0.35 to 2.04 mm per month, which is influenced by various factors and variables including the biological response of the individual to orthodontic forces, the complexity of the case, treatment mechanics and patient compliance throughout the course of treatment .

DETAILED DESCRIPTION:
To compare the alignment efficiency and pain experience of Mico-one self-ligating and conventional ligating MBT pre-adjusted brackets in the initial alignment stage of patients undergoing orthodontic treatment.CONVENTIONAL MBT BRACKETS: In conventional brackets elastic ligatures or metal ties are used to ligate the wire in the bracket slot. 2. SELF-LIGATING BRACKETS: Self-ligating brackets like conventional braces are placed relatively the same way.

The exception is that self-ligating braces don't use elastics, or metal ties. Instead it has special clips or brackets with a spring-loaded door. The brackets while maintaing pressure on the archwire, help move the teeth along it at a steady pace .[9] 3 .ALIGNMENT EFFICIENCY Movement of the teeth measured at four months interval. Scoring method involves measuring the linear distance between anatomical contact points between maxillary and mandibular incisors from adjacent tooth anatomical points. (Little's irregularity index)

4.PAIN Unpleasant sensory and emotional experience associated with tooth movement will be measured as a mean using the VAS at 4 hours, 24 hours, day 3, day 7, 1 st Month, 2 nd Month, 3 rd Month and 4 th Month.

ELIGIBILITY:
Inclusion Criteria

* Patients with Non extraction orthodontic treatment plan
* Crowding of 3 to 6 mm according to Little's irregularity index
* Both male and female patients
* 14-20 years of age.
* All permanent teeth present up to first permanent molar

Exclusion Criteria:

* Poor oral hygiene
* Systemic disease
* Patients with periodontally compromised teeth
* Patient requiring Orthognathic surgery to correct skeletal discrepancies
* Patients taking medications, like NSAIDs or other anti-inflammatory drugs
* Cleft lip or palate
* Hypodontia, or Hyperdontia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Alignment efficiency | 4 months
  amount of tooth movement in millimeters

SECONDARY OUTCOMES:
Pain with tooth movement | Four months
  pain perception using visual analogue scale with Zero equivalent to no pain and 10 indicates the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Zainab Butt, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No
To compare the alignment efficiency and pain experience of Mico-one self-ligating and conventional ligating MBT pre-adjusted brackets in the initial alignment stage of patients undergoing orthodontic treatment.

REFERENCES:
- [Background] 1. Wagner D, Lévy-Benichou H, Lefebvre F, Bolender Y. [Are self-ligating brackets more efficient than conventional brackets ? A meta-analysis of randomized controlled and split-mouth trials]. L' Orthodontie Francaise. 2020 Dec;91(4):303-321 2. Tantidhnazet S, Leehathorn P, Rattanasumawong S, Santiwong P. Comparison of self-ligating bracket and conventional bracket in orthodontic treatment: A systematic review. M Dent J 2018; 38: 213-228 3. Dehbi H, Azaroual MF, Zaoui F, Halimi A, Benyahia H. Therapeutic efficacy of self-ligating brackets: A systematic review. Int Orthod. 2017 Sep;15(3):297-311. 4. Jahanbin A, Hasanzadeh N, Khaki S, Shafaee H. Comparison of self-ligating Damon3 and conventional MBT brackets regarding alignment efficiency and pain experience: A randomized clinical trial. J Dent Res Dent Clin Dent Prospects. 2019 Fall;13(4):281-288. 5. Galvão MCS, Sato JR, Coelho EC. Dahlberg formula - a novel approach for its evaluation. Dental Press J Orthod. 2012;17(1):115-24.)